CLINICAL TRIAL: NCT00870623
Title: Procalcitonin and Endotoxin Sequential Levels to Optimize the Treatment of Bloodstream Infections
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0540-08-FB
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Bloodstream Infection
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood (maximum 40mL) will be collected for future use or for purposes that are not integral to the current research.
Oversight: Data Monitoring Committee: No

SUMMARY:
Bloodstream infections (BSI) are a major cause of morbidity and mortality. Bloodstream infections are also costly and result in prolonged hospital stays. The duration of therapy necessary to clear blood stream infections is unknown and no study has systematically addressed this issue. However, the use of antimicrobials is not without consequence. These include financial cost, side-effects, promotion of superinfection (especially Clostridium difficile-associated diarrhea), and the promotion of microbial resistance. This study hypothesizes that a procalcitonin (host biomarker) and endotoxin (microorganism biomarker) guided treatment plan could significantly decrease unnecessary exposure to antibiotics in patients with bloodstream infections.

DETAILED DESCRIPTION:
Bloodstream infections (BSI) are a major cause of morbidity and mortality. Community-onset BSI have an overall attributable mortality of 10-13% while nosocomial BSI mortality ranges are quite variable from 12-80%. Bloodstream infections are also costly and result in prolonged hospital stays. Nosocomial BSIs have been shown to increase length of stay by 5-25 days and increase costs $23,000 - 40,000 above matched controls. The duration of therapy necessary to clear blood stream infections is unknown and no study has systematically addressed this issue. The use of antimicrobials is also not without consequence. These include financial cost, side-effects, promotion of superinfection (especially Clostridium difficile-associated diarrhea), and the promotion of microbial resistance. This study hypothesizes that a procalcitonin (host biomarker) and endotoxin (microorganism biomarker) guided treatment plan could significantly decrease unnecessary exposure to antibiotics in patients with bloodstream infections.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized, adult patient, at least one positive blood culture reported within 24 hours of enrollment

Exclusion Criteria:

* Previously enrolled in the study; discharged/deceased before first positive culture; receiving antibiotic for greater than or equal to 48 hours; endocarditis or osteomyelitis; antithymocyte globulin in the last 12 months; blood cultures positive for coagulase-negative staphylococcus only.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized adult patients with positive blood cultures
Sampling Method: Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2009-06-01 (Actual); Primary Completion 2016-01-13 (Actual); Study Completion 2016-01-13 (Actual)

PRIMARY OUTCOMES:
Optimal length of treatment | 30 days
  To determine the optimal length of treatment by observing the normalization of procalcitonin (PCT) and Endotoxin levels, compared with the length of treatment by standard of care.

SECONDARY OUTCOMES:
Association of procalcitonin and endotoxin levels and outcomes | 30 days
  To determine if procalcitonin and endotoxin levels (or lack of decrease) are associated with treatment failure, complication, survival, cost, length of stay, progression to severe sepsis, or superinfections.

CONTACTS AND LOCATIONS:
Overall Officials: Andre Kalil, MD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] Diekema DJ, Beekmann SE, Chapin KC, Morel KA, Munson E, Doern GV. Epidemiology and outcome of nosocomial and community-onset bloodstream infection. J Clin Microbiol. 2003 Aug;41(8):3655-60. doi: 10.1128/JCM.41.8.3655-3660.2003. PMID 12904371
- [Background] Wisplinghoff H, Bischoff T, Tallent SM, Seifert H, Wenzel RP, Edmond MB. Nosocomial bloodstream infections in US hospitals: analysis of 24,179 cases from a prospective nationwide surveillance study. Clin Infect Dis. 2004 Aug 1;39(3):309-17. doi: 10.1086/421946. Epub 2004 Jul 15. PMID 15306996
- [Background] Laupland KB, Gregson DB, Flemons WW, Hawkins D, Ross T, Church DL. Burden of community-onset bloodstream infection: a population-based assessment. Epidemiol Infect. 2007 Aug;135(6):1037-42. doi: 10.1017/S0950268806007631. Epub 2006 Dec 7. PMID 17156500
- [Background] Shorr AF, Tabak YP, Killian AD, Gupta V, Liu LZ, Kollef MH. Healthcare-associated bloodstream infection: A distinct entity? Insights from a large U.S. database. Crit Care Med. 2006 Oct;34(10):2588-95. doi: 10.1097/01.CCM.0000239121.09533.09. PMID 16915117
- [Background] Digiovine B, Chenoweth C, Watts C, Higgins M. The attributable mortality and costs of primary nosocomial bloodstream infections in the intensive care unit. Am J Respir Crit Care Med. 1999 Sep;160(3):976-81. doi: 10.1164/ajrccm.160.3.9808145. PMID 10471627
- [Background] Warren DK, Quadir WW, Hollenbeak CS, Elward AM, Cox MJ, Fraser VJ. Attributable cost of catheter-associated bloodstream infections among intensive care patients in a nonteaching hospital. Crit Care Med. 2006 Aug;34(8):2084-9. doi: 10.1097/01.CCM.0000227648.15804.2D. PMID 16763511
- [Background] Pittet D, Tarara D, Wenzel RP. Nosocomial bloodstream infection in critically ill patients. Excess length of stay, extra costs, and attributable mortality. JAMA. 1994 May 25;271(20):1598-601. doi: 10.1001/jama.271.20.1598. PMID 8182812
- [Background] Mermel LA, Farr BM, Sherertz RJ, Raad II, O'Grady N, Harris JS, Craven DE; Infectious Diseases Society of America; American College of Critical Care Medicine; Society for Healthcare Epidemiology of America. Guidelines for the management of intravascular catheter-related infections. Clin Infect Dis. 2001 May 1;32(9):1249-72. doi: 10.1086/320001. Epub 2001 Apr 3. No abstract available. PMID 11303260
- [Background] Mandell LA, Wunderink RG, Anzueto A, Bartlett JG, Campbell GD, Dean NC, Dowell SF, File TM Jr, Musher DM, Niederman MS, Torres A, Whitney CG; Infectious Diseases Society of America; American Thoracic Society. Infectious Diseases Society of America/American Thoracic Society consensus guidelines on the management of community-acquired pneumonia in adults. Clin Infect Dis. 2007 Mar 1;44 Suppl 2(Suppl 2):S27-72. doi: 10.1086/511159. No abstract available. PMID 17278083
- [Background] Warren JW, Abrutyn E, Hebel JR, Johnson JR, Schaeffer AJ, Stamm WE. Guidelines for antimicrobial treatment of uncomplicated acute bacterial cystitis and acute pyelonephritis in women. Infectious Diseases Society of America (IDSA). Clin Infect Dis. 1999 Oct;29(4):745-58. doi: 10.1086/520427. PMID 10589881
- [Background] Corona A, Bertolini G, Ricotta AM, Wilson A, Singer M. Variability of treatment duration for bacteraemia in the critically ill: a multinational survey. J Antimicrob Chemother. 2003 Nov;52(5):849-52. doi: 10.1093/jac/dkg447. Epub 2003 Sep 30. PMID 14519681
- [Background] Corona A, Wilson AP, Grassi M, Singer M. Prospective audit of bacteraemia management in a university hospital ICU using a general strategy of short-course monotherapy. J Antimicrob Chemother. 2004 Oct;54(4):809-17. doi: 10.1093/jac/dkh416. Epub 2004 Sep 16. PMID 15375106
- [Background] Rice LB. The Maxwell Finland Lecture: for the duration-rational antibiotic administration in an era of antimicrobial resistance and clostridium difficile. Clin Infect Dis. 2008 Feb 15;46(4):491-6. doi: 10.1086/526535. PMID 18194098
- [Background] Christ-Crain M, Jaccard-Stolz D, Bingisser R, Gencay MM, Huber PR, Tamm M, Muller B. Effect of procalcitonin-guided treatment on antibiotic use and outcome in lower respiratory tract infections: cluster-randomised, single-blinded intervention trial. Lancet. 2004 Feb 21;363(9409):600-7. doi: 10.1016/S0140-6736(04)15591-8. PMID 14987884
- [Background] Christ-Crain M, Stolz D, Bingisser R, Muller C, Miedinger D, Huber PR, Zimmerli W, Harbarth S, Tamm M, Muller B. Procalcitonin guidance of antibiotic therapy in community-acquired pneumonia: a randomized trial. Am J Respir Crit Care Med. 2006 Jul 1;174(1):84-93. doi: 10.1164/rccm.200512-1922OC. Epub 2006 Apr 7. PMID 16603606
- [Background] Stolz D, Christ-Crain M, Bingisser R, Leuppi J, Miedinger D, Muller C, Huber P, Muller B, Tamm M. Antibiotic treatment of exacerbations of COPD: a randomized, controlled trial comparing procalcitonin-guidance with standard therapy. Chest. 2007 Jan;131(1):9-19. doi: 10.1378/chest.06-1500. PMID 17218551
- [Background] Nobre V, Harbarth S, Graf JD, Rohner P, Pugin J. Use of procalcitonin to shorten antibiotic treatment duration in septic patients: a randomized trial. Am J Respir Crit Care Med. 2008 Mar 1;177(5):498-505. doi: 10.1164/rccm.200708-1238OC. Epub 2007 Dec 20. PMID 18096708
- [Background] Tang BM, Eslick GD, Craig JC, McLean AS. Accuracy of procalcitonin for sepsis diagnosis in critically ill patients: systematic review and meta-analysis. Lancet Infect Dis. 2007 Mar;7(3):210-7. doi: 10.1016/S1473-3099(07)70052-X. PMID 17317602
- [Background] Giamarellos-Bourboulis EJ, Grecka P, Poulakou G, Anargyrou K, Katsilambros N, Giamarellou H. Assessment of procalcitonin as a diagnostic marker of underlying infection in patients with febrile neutropenia. Clin Infect Dis. 2001 Jun 15;32(12):1718-25. doi: 10.1086/320744. Epub 2001 May 21. PMID 11360214
- [Background] Jensen JU, Heslet L, Jensen TH, Espersen K, Steffensen P, Tvede M. Procalcitonin increase in early identification of critically ill patients at high risk of mortality. Crit Care Med. 2006 Oct;34(10):2596-602. doi: 10.1097/01.CCM.0000239116.01855.61. PMID 16915118
- [Background] Romaschin AD, Harris DM, Ribeiro MB, Paice J, Foster DM, Walker PM, Marshall JC. A rapid assay of endotoxin in whole blood using autologous neutrophil dependent chemiluminescence. J Immunol Methods. 1998 Mar 15;212(2):169-85. doi: 10.1016/s0022-1759(98)00003-9. PMID 9672205
- [Background] Marshall JC, Walker PM, Foster DM, Harris D, Ribeiro M, Paice J, Romaschin AD, Derzko AN. Measurement of endotoxin activity in critically ill patients using whole blood neutrophil dependent chemiluminescence. Crit Care. 2002 Aug;6(4):342-8. doi: 10.1186/cc1522. Epub 2002 May 2. PMID 12225611
- [Background] Marshall JC, Foster D, Vincent JL, Cook DJ, Cohen J, Dellinger RP, Opal S, Abraham E, Brett SJ, Smith T, Mehta S, Derzko A, Romaschin A; MEDIC study. Diagnostic and prognostic implications of endotoxemia in critical illness: results of the MEDIC study. J Infect Dis. 2004 Aug 1;190(3):527-34. doi: 10.1086/422254. Epub 2004 Jul 2. PMID 15243928
- [Background] Bates DW, Cullen DJ, Laird N, Petersen LA, Small SD, Servi D, Laffel G, Sweitzer BJ, Shea BF, Hallisey R, et al. Incidence of adverse drug events and potential adverse drug events. Implications for prevention. ADE Prevention Study Group. JAMA. 1995 Jul 5;274(1):29-34. PMID 7791255
- [Background] McFarland LV, Clarridge JE, Beneda HW, Raugi GJ. Fluoroquinolone use and risk factors for Clostridium difficile-associated disease within a Veterans Administration health care system. Clin Infect Dis. 2007 Nov 1;45(9):1141-51. doi: 10.1086/522187. Epub 2007 Sep 26. PMID 17918075
- [Background] Chastre J, Wolff M, Fagon JY, Chevret S, Thomas F, Wermert D, Clementi E, Gonzalez J, Jusserand D, Asfar P, Perrin D, Fieux F, Aubas S; PneumA Trial Group. Comparison of 8 vs 15 days of antibiotic therapy for ventilator-associated pneumonia in adults: a randomized trial. JAMA. 2003 Nov 19;290(19):2588-98. doi: 10.1001/jama.290.19.2588. PMID 14625336